CLINICAL TRIAL: NCT04973878
Title: The Optimal Sequence in Same-day Bidirectional Endoscopy Under Deep Anesthesia Induced by Propofol Combined With Fentanyl: A Prospective Randomized Controlled ,Two Centers Trial
Brief Title: The Optimal Sequence in Same-day Bidirectional Endoscopy Under Deep Anesthesia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, duowu zou, prof. and director, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RuijinH2021131
Record Dates: First submitted 2021-07-17; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Bidirectional Endoscopy; Deep Sedation
Keywords: Bidirectional Endoscopy; Deep Sedation

STUDY DESIGN:
Intervention Model Description: Patients undergoing same-day bidirectional endoscopy under deep sedation will be randomly assigned to either the colonoscopy-first group (colonoscopy followed by EGD, n = 272) or the EGD-first group (EGD followed by colonoscopy, n = 272).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): EGD performed before the Colonoscopy
  Interventions: Procedure: EGD first
- Group B (Experimental): Colonoscopy performed before the EGD
  Interventions: Procedure: Colonoscopy first

INTERVENTIONS:
Procedure: EGD first — In this group, patients receiving an EGD followed by a colonoscopy during a same-day bidirectional endoscopy. Patients receive deep sedation with propofol and fentanyl.
  Arms: Group A
Procedure: Colonoscopy first — In this group, patients receiving a colonoscopy followed by EGD during a same-day bidirectional endoscopy. Patients receive deep sedation with propofol and fentanyl.
  Arms: Group B

SUMMARY:
The purpose of this study is to explore the optimal sequence of same-day bidirectional endoscopy under deep anesthesia induced by propofol combined with fentanyl.

DETAILED DESCRIPTION:
Same-day bidirectional endoscopy are commonly performed to evaluate iron deficiency anemia, positive fecal occult blood, abdominal pain and cancer screening. In order to reducing intraoperative pain, providing better operating conditions and improving the endoscopic examination quality, endoscopy with anesthesia assistance has gradually become the choice of more patients. However, the optimal sequence of procedures for same-day bidirectional endoscopy has not been established. This is a two-center, single-blind, randomized, controlled trial. Patients undergoing same-day bidirectional endoscopy under deep sedation will be randomly assigned to either the colonoscopy-first group (colonoscopy followed by EGD, n = 272) or the EGD(esophagogastroduodenoscopy)-first group (EGD followed by colonoscopy, n = 272).The detection rate of adenoma（ADR）, the ADR of right-side colon , Boston score of right-side colon, total dose of anesthetics, operation time, recovery time, adverse events and patient satisfaction will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a clinical indication for receiving same day bi-directional endoscopies.

Exclusion Criteria:

* Contraindications of colonoscopy: acute peritonitis; intestinal perforation or suspected intestinal perforation; acute anorectal infection or painful lesions; menstruation; pregnancy; cardiopulmonary insufficiency; prior abdominal and pelvic surgery.
* Contraindications for EGD: severe heart disease, severe heart failure; severe lung disease: asthma : severe hypertension; acute perforation of esophagus, stomach and duodenum; acute severe pharynx and larynx disease gastroscopy can not be inserted; acute stage of corrosive esophageal injury; prior upper digestive tract operation.
* Contraindications for oral intestinal laxative: severe gastrointestinal obstruction or stricture; toxic megacolon; severe acute intestinal infection; dysphagia; disturbance of consciousness; allergy to drug ingredients.
* Allergic to emulsions or opioids.
* ASA score ≥ III

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 544 (Estimated)
Dates: Start 2021-07-30 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Adenoma Detection Rate | 1 year
  Adenoma detection rate is the proportion of individuals undergoing a complete screening colonoscopy who have one or more adenomas detected. In this study, ADR during the colonoscopy will recorded.
Adenoma Detection Rate of the right-sided colon | 1 year
  The ADR of right-sided colon will be recorded.Right -sided colon is refered to cecum, ascending colon and ileocecal junction.
The boston bowel preparation scale of the right-sided colon | 1 year
  During colonoscopy, the boston bowel preparation scale of the right-sided colon will be recorded and compared between the two study groups.

SECONDARY OUTCOMES:
Sedation use | 1 year
  During bidirectional endoscopy, the total doses of propofol and fentanyl will be recorded.
Overall Duration of BDE Examinations | 1 year
  The overall duration of both EGD and colonoscopy examinations will be recorded.
Recovery time | 1 year
  Time between the end of the procedure and patient waken-up will be recorded.
Adverse events | 1 year
  Intraprocedure adverse events will be documented (oxygen saturation <90% for >30 s, systolic blood pressure drop for 30 %, and heart rate <50 or >120 beats/min lasting >30 s).
Overall patient satisfaction | 1 year
  Patient satisfaction will be assessed after the procedures using 10-cm visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Duowu Zou, Ph.D,M.D, Study Chair — Ruijin hospital Shanghai Jiaotong Universtity, school of medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Urquhart J, Eisen G, Faigel DO, Mattek N, Holub J, Lieberman DA. A closer look at same-day bidirectional endoscopy. Gastrointest Endosc. 2009 Feb;69(2):271-7. doi: 10.1016/j.gie.2008.04.063. Epub 2008 Aug 23. PMID 18725159
- [Background] Cairns SR, Scholefield JH, Steele RJ, Dunlop MG, Thomas HJ, Evans GD, Eaden JA, Rutter MD, Atkin WP, Saunders BP, Lucassen A, Jenkins P, Fairclough PD, Woodhouse CR; British Society of Gastroenterology; Association of Coloproctology for Great Britain and Ireland. Guidelines for colorectal cancer screening and surveillance in moderate and high risk groups (update from 2002). Gut. 2010 May;59(5):666-89. doi: 10.1136/gut.2009.179804. PMID 20427401
- [Background] Lucendo AJ, Arias A, Gonzalez-Castillo S, Angueira T, Guagnozzi D, Fernandez-Fuente M, Serrano-Valverde M, Sanchez-Cazalilla M, Chumillas O, Fernandez-Ordonez M, Tenias JM. Same-day bidirectional endoscopy with nonanesthesiologist administration of propofol: safety and cost-effectiveness compared with separated exams. Eur J Gastroenterol Hepatol. 2014 Mar;26(3):301-8. doi: 10.1097/MEG.0000000000000026. PMID 24365718
- [Background] Yang C, Sriranjan V, Abou-Setta AM, Poluha W, Walker JR, Singh H. Anxiety Associated with Colonoscopy and Flexible Sigmoidoscopy: A Systematic Review. Am J Gastroenterol. 2018 Dec;113(12):1810-1818. doi: 10.1038/s41395-018-0398-8. Epub 2018 Nov 1. PMID 30385831
- [Background] Lu Y, Hao LX, Chen L, Jin Z, Gong B. Systematic review and meta-analysis of patient-controlled sedation versus intravenous sedation for colonoscopy. Int J Clin Exp Med. 2015 Nov 15;8(11):19793-803. eCollection 2015. PMID 26884890
- [Background] Igea F, Casellas JA, Gonzalez-Huix F, Gomez-Oliva C, Baudet JS, Cacho G, Simon MA, De la Morena E, Lucendo A, Vida F; Spanish Society of Digestive Endoscopy. Sedation for gastrointestinal endoscopy. Endoscopy. 2014 Aug;46(8):720-31. doi: 10.1055/s-0034-1377561. Epub 2014 Jul 25. No abstract available. PMID 25061964
- [Background] Bugajski M, Wieszczy P, Hoff G, Rupinski M, Regula J, Kaminski MF. Modifiable factors associated with patient-reported pain during and after screening colonoscopy. Gut. 2018 Nov;67(11):1958-1964. doi: 10.1136/gutjnl-2017-313905. Epub 2017 Sep 28. PMID 28970289
- [Background] Grocott HP. Propofol sedation improves efficiency and optimizes patient satisfaction during colonoscopy. CMAJ. 2018 Jun 18;190(24):E751. doi: 10.1503/cmaj.69279. No abstract available. PMID 29914915
- [Background] Wadhwa V, Issa D, Garg S, Lopez R, Sanaka MR, Vargo JJ. Similar Risk of Cardiopulmonary Adverse Events Between Propofol and Traditional Anesthesia for Gastrointestinal Endoscopy: A Systematic Review and Meta-analysis. Clin Gastroenterol Hepatol. 2017 Feb;15(2):194-206. doi: 10.1016/j.cgh.2016.07.013. Epub 2016 Jul 21. PMID 27451091
- [Background] Cao Y, Yang J, Li J, Ao X, Zhang KY, Shen XC, Chen DF, Lan CH. Comparison of procedural sequences in same-day painless bidirectional endoscopy: Single-center, prospective, randomized study. Dig Endosc. 2017 May;29(3):330-337. doi: 10.1111/den.12847. Epub 2017 Mar 30. PMID 28211094
- [Background] Hsieh YH, Lin HJ, Tseng KC. Which should go first during same-day bidirectional endosocopy with propofol sedation? J Gastroenterol Hepatol. 2011 Oct;26(10):1559-64. doi: 10.1111/j.1440-1746.2011.06786.x. PMID 21615790
- [Background] Hammami MB, Reddy KM, Pandit P, Chahla EJ, Koro N, Schuelke MJ, Hachem C. Sequence of same-day upper and lower gastrointestinal endoscopy does not affect total procedure' time or medication use: A randomized trial. JGH Open. 2019 Aug 6;3(6):488-493. doi: 10.1002/jgh3.12203. eCollection 2019 Dec. PMID 31832549
- [Background] Rex DK, Schoenfeld PS, Cohen J, Pike IM, Adler DG, Fennerty MB, Lieb JG 2nd, Park WG, Rizk MK, Sawhney MS, Shaheen NJ, Wani S, Weinberg DS. Quality indicators for colonoscopy. Gastrointest Endosc. 2015 Jan;81(1):31-53. doi: 10.1016/j.gie.2014.07.058. Epub 2014 Dec 2. No abstract available. PMID 25480100
- [Background] Chokshi RV, Hovis CE, Hollander T, Early DS, Wang JS. Prevalence of missed adenomas in patients with inadequate bowel preparation on screening colonoscopy. Gastrointest Endosc. 2012 Jun;75(6):1197-203. doi: 10.1016/j.gie.2012.01.005. Epub 2012 Feb 28. PMID 22381531